CLINICAL TRIAL: NCT02239887
Title: Coherex WAVECREST I Left Atrial Appendage Occlusion Study
Status: Completed | Type: Observational
Sponsor: Coherex Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: IP005
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Non-valvular Paroxysmal, Persistent, or Permanent Atrial Fibrillation; LAA Anatomy Amenable to Treatment by Percutaneous Technique; Anticoagulation Indication for Potential Thrombus Formation in the Left Atrium
Keywords: LAA occlusion; Non-valvular Atrial Fibrillation; Percutaneous; Oral Anticoagulation; Occluder; WAVECREST

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- WaveCrest LAA occlusion device: Left Atrial Occlusion
  Interventions: Device: WaveCrest LAA occlusion device

INTERVENTIONS:
Device: WaveCrest LAA occlusion device — Left Atrial Appendage Occlusion

SUMMARY:
Purpose To establish the safety and efficacy of the Coherex WaveCrest Left Atrial Appendage Occlusion System for left atrial appendage (LAA) closure during treatment of non-valvular atrial fibrillation in patients who are at increased risk for embolic stroke and have an ongoing indication for oral anticoagulation.

DETAILED DESCRIPTION:
Primary Safety Endpoint The primary safety endpoint is the incidence of major adverse events up to 45 days post-procedure. Major adverse events are defined as life-threatening incidents as determined by the Clinical Events Committee (CEC) and include events such as device embolization; cardiac injury, re-intervention, and/or device-related surgery; bleeding events such as pericardial effusion requiring drainage, cranial bleeding due to any source, gastrointestinal bleeding; or any other event related to the device or the procedure, which requires treatment.

Primary Efficacy Endpoint The primary efficacy endpoint is the incidence of LAA occlusion at 45 and/or 180 days (+ten days) post-procedure. LAA occlusion will be assessed by transesophageal echocardiography (TEE) color flow Doppler and will be defined as absence of flow in the LAA or color flow Doppler jets less than 3mm.

ELIGIBILITY:
Inclusion Criteria:Candidates for this study must meet ALL of the following criteria

1. At least 18 years of age.
2. Diagnosis of paroxysmal, persistent, or permanent non-valvular atrial fibrillation.
3. Indicated for long-term anticoagulation therapy including patients on anticoagulants and patients with a contraindication to anticoagulation. The first 30 patients must have a contraindication to anticoagulation.
4. Eligible for cessation of anticoagulation therapy if the LAA is sealed (i.e., the patient has no other condition requiring anticoagulation therapy).
5. Calculated CHADS score ≥ 1.
6. Willingness to participate in the required follow-up visits and tests.
7. Willingness of patient or legal representative to provide written informed consent.
8. Female subjects of child-bearing potential must have a negative serum pregnancy test within 7 days prior to the index procedure, and must be willing to use reliable contraception methods for one year post-procedure.

Exclusion Criteria:

1. Known contraindication and/or allergy to aspirin, clopidogrel, IV contrast, or nickel.
2. Extensive congenital cardiac anomalies, which can only be adequately repaired by cardiac surgery.
3. Stroke or transient ischemic attack (TIA), as diagnosed by a neurologist, within the past 30 days. Patients with a history of stroke or TIA will not be allowed to enroll until 30 days post stroke or TIA have been completed.
4. New York Heart Association Class IV Congestive Heart Failure, defined as patients with severe physical limitations and symptoms even while at rest.
5. Myocardial infarction within the past three months.
6. Sepsis within one month prior to implantation or any systemic infection that cannot be successfully treated prior to device placement.
7. Presence of an atrial septal defect, atrial septal repair, or atrial septal closure device.
8. Female subjects who may be pregnant or are planning on becoming pregnant in the next year.
9. Cardioversion or ablation procedure planned in conjunction with or within 30 days after placement of the Coherex WaveCrest Left Atrial Appendage Occlusion System.
10. Cardiac transplant or mechanical valve.
11. Symptomatic carotid artery disease.
12. Any medical disorder or psychiatric illness that would interfere with successful completion of the study as determined by the investigator.
13. Conditions other than atrial fibrillation requiring long-term warfarin therapy.
14. Resting heart rate > 110 beats per minute (bpm).
15. A single episode of transient atrial fibrillation.
16. Thrombocytopenia (<50,000 platelets/mm3), thrombocythemia (>700,000 platelets/mm³), leucopenia (white blood cell count < 3,000 cells/mm³), or anemia (hemoglobin concentration < 10 gram per deciliter [g/dl]).
17. Currently participating in an investigational drug or another device trial that has not completed the primary endpoint or that clinically interferes with the current trial endpoints. (Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials.)
18. Any condition that would reduce life expectancy to less than two years from the date of the index procedure.

Echocardiographic criteria for exclusion:

1. Left ventricular ejection fraction (LVEF) < 30%.
2. Mitral valve stenosis < 1.5 cm2 or any stenosis consistent with rheumatic valvular disease.
3. Pericardial effusion > 5 mm pre-procedure.
4. Evidence of intracardiac thrombus visualized on TEE.
5. Presence of a patent foramen ovale (PFO) that demonstrates a large shunt and/or atrial septal aneurysm with > 10 mm excursion.
6. Cardiac tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population for this study is the subset of patients who have non-valvular paroxysmal, persistent, or permanent atrial fibrillation; LAA anatomy amenable to treatment by percutaneous techniques; and an anticoagulation indication for potential thrombus formation in the left atrium. Patients with an absolute or relative contraindication to anticoagulants will also be included.
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2010-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint | 45 Days post procedure
  The primary safety endpoint is the incidence of major adverse events up to 45 days post-procedure. Major adverse events are defined as life-threatening incidents as determined by the Clinical Events Committee (CEC) and include events such as device embolization; cardiac injury, re-intervention, and/or device-related surgery; bleeding events such as pericardial effusion requiring drainage, cranial bleeding due to any source, gastrointestinal bleeding; or any other event related to the device or the procedure, which requires treatment.
Primary Efficacy Endpoint | 45 and/or 180 days post procedure
  The primary efficacy endpoint is the incidence of LAA occlusion at 45 and/or 180 days (+ten days) post-procedure. LAA occlusion will be assessed by transesophageal echocardiography (TEE) color flow Doppler and will be defined as absence of flow in the LAA or color flow Doppler jets less than 3mm.

SECONDARY OUTCOMES:
Secondary Safety Endpoint | 180 days and one year post-procedure
  The secondary safety endpoint is the incidence of serious adverse events at 180 days and one year post-procedure. Serious adverse events are defined as any events that result in death, are life-threatening, require in-patient hospitalization or prolongation of existing hospitalization, or result in permanent or significant disability/incapacity.
Secondary Efficacy Endpoints | intra operative
  1. Procedural success, defined as successful delivery, deployment, and release of the Coherex WaveCrest Left Atrial Appendage Occlusion System into the LAA, and includes successful recapture and retrieval, if necessary.
  2. The incidence of LAA occlusion as measured by echocardiographic color flow Doppler jets less than 3mm by TEE at the end of the procedure.